CLINICAL TRIAL: NCT05695859
Title: SPECT/CT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Primary Tumour and Metastatic Axillary Lymph Nodes Using Technetium-99m-labelled DARPinG3 Molecule-based.
Brief Title: 99mTc-DARPinG3 SPECT/CT for Non-invasive HER2-AX in Breast Cancer With Metastatic Lymph Nodes Before Targeted Therapy
Status: Completed | Type: Observational
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 99mTc-DARPinG3 breast cancer
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer Female
Keywords: 99mTc-DARPinG3; breast cancer; metastatic lymph nodes; HER2
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: 99mTc-DARPinG3 SPECT/CT — One single injection of 99mTc-DARPinG3, followed by gamma camera imaging 4 hours after injection
  Other Names: SPECT/CT

SUMMARY:
An open-label, single center study with 99mTc-DARPinG3 SPECT/CT and biopsies of primary tumour and metastatic lymph nodes in breast cancer patients, where the primary endpoint of the study is to find out the correlation between the HER2 expression measured by 99mTc-DARPinG3 SPECT/CT and standard histopathology from relevant tumor and lymph node biopsies.

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer and axillary lymph node metastases before chemo/targeted therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Diagnosis of primary breast cancer with lymph node metastases
* Availability of results from HER2 status previously determined on material from the primary tumor and metastatic LN, either a. HER2-positive, defined as a DAKO HercepTest™ score of 3+ or FISH positive or b. HER2-negative, defined as a DAKO HercepTest™ score of 0 or 1+; or else if 2+ then FISH negative
* Hematological, liver and renal function test results within the following limits: White blood cell count: > 2.0 x 109/L; Hemoglobin: > 80 g/L; Platelets: > 50.0 x 109/L; ALT, ALP, AST: =< 5.0 times Upper Limit of Normal; Bilirubin =< 2.0 times Upper Limit of Normal; Serum creatinine: Within Normal Limits.
* A negative pregnancy test for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Any system therapy (chemo-/targeted therapy)
* Second, non-breast malignancy
* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening) 4. Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer female patients
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
SPECT/CT-based 99mTc-DARPinG3 uptake in tumor lesions | 4 hours
  SPECT/CT-based 99mTc-DARPinG3 uptake value in tumor lesions (counts)/SUV of 99mTc-DARPinG3 focal uptake coinciding with tumor lesions is assessed using SPECT/CT at 4 hours after injection and measured in counts and SUV
SPECT/CT-based 99mTc-DARPinG3 uptake value in metastatic lymph nodes | 4 hours
  SPECT/CT-based 99mTc-DARPinG3 uptake value in metastatic lymph nodes (counts)/SUV of 99mTc-DARPinG3 focal uptake coinciding with tumor lesions is assessed using SPECT/CT at 4 hours after injection and measured in counts and SUV
Tumor-to-background ratio (SPECT) | 4 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-DARPinG3 uptake coinciding with tumor lesions (counts/SUV) will be divided by the value of 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (counts/SUV)
LN-to-background LN ratio (SPECT) | 4 hours
  The SPECT-based LN-to-background LN ratio will be calculated as follows: the value of 99mTc-DARPinG3 uptake coinciding with LN lesions (counts/SUV) will be divided by the value of 99mTc-DARPinG3 uptake coinciding with the regions without pathological findings (counts/SUV)

SECONDARY OUTCOMES:
Morphological and immunohistochemical verification of 99mTc-DARPinG3 accumulation | 4 hours
  Comparison of the 99mTc-DARPinG3 accumulation in the primary tumor and metastatic lymph nodes with the results of morphological and immunohistochemical studies

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Chernov, MD, Principal Investigator — Tomsk NRMC
Locations (1):
- Russia Tomsk NRMC, Tomsk, Russia